CLINICAL TRIAL: NCT00458068
Title: Prospective Randomized Trial of Early Versus Late Enteral Iron Supplementation in Infants With a Birth Weight of Less Than 1301 Grams
Brief Title: Early Versus Late Enteral Iron in Infants Less Than 1301 Grams
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: UL-NEO-IRON-1
Record Dates: First submitted 2007-04-06; First posted 2007-04-09 (Estimated); Last update posted 2007-04-09 (Estimated); Status verified 2007-04

CONDITIONS: Iron Deficiency; Anemia of Prematurity
Keywords: preterm infant; iron supplementation; iron deficiency; blood transfusion
MeSH Terms: conditions — Iron Deficiencies; Anemia; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Oral administration of ferrous sulphate

SUMMARY:
Background: Preterm infants are at risk of iron deficiency. The smaller the infants are at birth, the smaller the iron stores at birth and the higher the risk of iron deficiency.

Hypothesis: Preterm infants with a birth weight of less than 1301g require iron supplementation earlier than previously recommended.

Methods: Prospective randomized controlled clinical trial (1996-1999). Results: Early iron supplementation may reduce the incidence of iron deficiency and the need for late blood transfusions.

DETAILED DESCRIPTION:
Objectives. To examine whether early enteral iron supplementation (EI) would improve serum ferritin as a measure of nutritional iron status at 2 months of age and would prevent definite iron deficiency (ID) in infants with a birth weight of <1301 g. Methods. Infants were randomly assigned to receive enteral iron supplementation of 2 to 6 mg/kg/day as soon as enteral feedings of >100 mL/kg/day were tolerated (EI) or at 61 days of life (late enteral iron supplementation [LI]). Nutritional iron status was assessed: 1) at birth, 2) at 61 days of life, 3) when the infants reached a weight of 1.6 times birth weight, and 4) before blood was transfused at a hematocrit of <.25. ID was defined by any one of the following criteria: ferritin, <12 mg/L; transferrin saturation, <17%; or increase of absolute reticulocyte counts by >50% one week after the onset of enteral iron supplementation. Restrictive red cell transfusion guidelines were followed and all transfusions were documented. Erythropoietin was not administered. The primary outcome variables were: 1) ferritin at 61 days and 2) the number of infants with ID. Results. Ferritin at 61 days was not different between the groups. Infants in the LI group were more often iron-deficient (26/65 vs 10/68) and received more blood transfusions after day 14 of life. No adverse effects of EI were noted. Conclusions. EI is feasible and probably safe in infants with birth weight <1301 g. EI may reduce the incidence of ID and the number of late blood transfusions. ID may occur in very low birth weight infants despite early supplementation with iron and should be considered in the case of progressive anemia. Pediatrics 2000; 106:700 -706; preterm infant, iron supplementation, iron deficiency, blood transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Inborn infant
* Birth weight of <1301 g
* Admitted between June 1996 and June 1999

Exclusion Criteria:

* Major anomalies
* Hemolytic disease
* Twin-to-twin transfusion syndrome
* Missing parental consent

Ages: 3 Days to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126
Dates: Start 1996-06; Study Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
Ferritin at 61 days of life
The number of infants who fulfilled the criteria of ID at any time throughout the study.

SECONDARY OUTCOMES:
Transferrin-Saturation
Hematocrit at day 61
Reticulocyte count at day 61
Mean corpuscular volume at day 61
Mean corpuscular hemoglobin at day 61
Number of infants who required transfusions at days 14 to 68
Blood volume transfused at days 14 to 68

CONTACTS AND LOCATIONS:
Overall Officials: Axel R Franz, MD, Principal Investigator — University of Ulm
Locations (1):
- University Children's Hospital, Ulm, Germany

REFERENCES:
- [Result] Franz AR, Mihatsch WA, Sander S, Kron M, Pohlandt F. Prospective randomized trial of early versus late enteral iron supplementation in infants with a birth weight of less than 1301 grams. Pediatrics. 2000 Oct;106(4):700-6. doi: 10.1542/peds.106.4.700. PMID 11015511